CLINICAL TRIAL: NCT06862128
Title: Oral Glucose Tolerance Test at Home With Continuous Glucose Monitoring vs Standard Clinic-based Testing
Brief Title: OGTT at Home Using CGM vs at the Clinic
Acronym: OGTT-CGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Jönköping County (Other Government); Region Östergötland (Other)
Responsible Party: Principal Investigator, Peder af Geijerstam, Principal Investigator, Linkoeping University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ogtt_cgm
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pre-diabetes; Diabetes
Keywords: Pre-diabetes; Diabetes; Oral glucose tolerance test; Continuous glucose monitoring; Glucose
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OGTT at the clinic then at home (Experimental): OGTT at the clinic then at home
  Interventions: Diagnostic Test: OGTT at home using CGM; Diagnostic Test: OGTT at the clinic
- OGTT at home then at the clinic (Experimental): OGTT at home then at the clinic
  Interventions: Diagnostic Test: OGTT at home using CGM; Diagnostic Test: OGTT at the clinic

INTERVENTIONS:
Diagnostic Test: OGTT at home using CGM — OGTT at home using CGM
  Other Names: OGTT-home
Diagnostic Test: OGTT at the clinic — OGTT at the clinic
  Other Names: OGTT-clinic

SUMMARY:
This randomized, crossover study evaluates the feasibility and accuracy of a self-administered oral glucose tolerance test (OGTT) at home using continuous glucose monitoring (CGM) compared to a standard clinic-based OGTT. Participants with prediabetes will undergo both home-based and clinic-based OGTTs, with glucose levels measured via CGM and venous plasma glucose. The primary outcome is the correlation between CGM-based glucose values and standard OGTT results. Secondary outcomes include diagnostic agreement, metabolic hormone associations, and feasibility of home-based testing as a diagnostic tool for dysglycemia.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility, accuracy, and diagnostic utility of a self-administered oral glucose tolerance test (OGTT) at home using continuous glucose monitoring (CGM) compared to a standard clinic-based OGTT.

Study Design Type: Randomized, crossover study Participants: 75 adults with prediabetes Intervention: Each participant will complete both a home-based OGTT with CGM and a clinic-based OGTT with venous plasma glucose measurement.

Primary Objective To assess the correlation between glucose values obtained from a CGM-based home OGTT and a standard venous OGTT performed in the clinic.

Secondary Objectives Evaluate diagnostic agreement between CGM-derived and venous glucose measurements.

Assess variability in glucose responses between the two methods. Investigate associations between OGTT results and metabolic/sex hormones. Determine feasibility and patient adherence to home-based testing.

Methods Participants will be randomized into two groups: one starting with a clinic-based OGTT, the other with a home-based OGTT, followed by a crossover period. CGM will continuously monitor glucose responses, and standard venous plasma glucose measurements will serve as the reference method.

Clinical Relevance A validated home-based OGTT using CGM could improve access to glucose tolerance testing, reduce patient burden, and enhance early detection of dysglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes indicated by ≥2 of the following values, measured at separate occasions or through different analyses during the past 2 years:
* - Fasting venous plasma glucose ≥6.1 but ≤6.9 mmol/L
* - Non-fasting venous plasma glucose ≥7.8 but ≤11.0 mmol/L
* - HbA1c ≥39 but ≤47 mmol/mol
* Access to a smart phone which is compatible with the CGM application and has working Bluetooth connectivity
* Ability to read and respond to online instructions and questionnaires in Swedish.

Exclusion Criteria:

* T2D indicated by ≥2 of the following values, measured at different occasions or through different analyses:
* - Fasting venous plasma glucose ≥7.0 mmol/L
* - Non-fasting venous plasma glucose value ≥11.1 mmol/L
* - HbA1c ≥48 mmol/mol
* Previous bariatric surgery e.g., gastric by-pass or gastric sleeve surgery
* Body mass index <20 kg/m2
* Body weight <43 kg
* Current pregnancy
* Need of regular use of GLP-1 receptor agonists, SGLT-2 inhibitors, acetaminophen or ascorbic acid supplements during the study period
* Fear of needle sticks
* Shift work during the study period
* Involvement in the study design, data collection, analysis, or participant recruitment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
The correlation coefficient between the glucose levels of the OGTT-home vs OGTT-clinic | Between OGTT-clinic at baseline vs OGTT-home at each 5-min interval from 0-30 min; Between OGTT-clinic at 1 h vs OGTT-home at each 5-min interval from 60-90 min; Between OGTT-clinic at 2 h vs OGTT-home at each 5-min interval from 120-150 min
  The correlation coefficient between the glucose levels of the OGTT at home vs at the clinic
The sensitivity and specificity, as well as the positive and negative predictive values of the OGTT at home vs the OGTT at the clinic | At 1 and 2 hours after the start of the OGTT
  The sensitivity and specificity, as well as the positive and negative predictive values of pre-diabetes and diabetes of the OGTT-CGM with the highest correlation coefficient to the OGTT-CLI, at 1 and 2 hours after the start of the OGTT

SECONDARY OUTCOMES:
The sensitivity, specificity, positive and negative predictive value of the highest OGTT-home vs OGTT-clinic | Any of the values from 5-minute intervals 0-150 minutes of OGTT-home vs OGTT-clinic at 1 and 2 hours, respectively
  The sensitivity, specificity, positive and negative predictive value of the highest glucose value form the OGTT at home vs the value of OGTT at the clinic at 1 and 2 hours, respectively
The sensitivity, specificity, positive and negative predictive value of the highest CGM value vs OGTT-clinic | Any of the values from 5-minute intervals days 1-14 of the CGM vs OGTT-clinic at 1 and 2 hours, respectively
  The sensitivity, specificity, positive and negative predictive value of the highest glucose value form the CGM vs the value of OGTT at the clinic at 1 and 2 hours, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Peder af Geijerstam, MD, PhD, Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - Primary Health Care Center Bra Liv Rosenhälsan, Huskvarna, Jönköping County
  - Primary Health Care Center Cityhälsan Centrum, Norrköping, Norrköping
  - Primary Care Center Vårdcentralen Kärna, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Undecided
If suitable according to ethical guidelines.